CLINICAL TRIAL: NCT06424067
Title: A Phase II Study of Fingolimod in Patients With Non-Small Cell and Small Cell Lung Cancer
Brief Title: Phase 2 Study of Fingolimod in Lung Cancers
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Mariam Alexander, Assistant Professor-Faculty, Medical University of South Carolina
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 103909
Record Dates: First submitted 2024-04-18; First posted 2024-05-21 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-04

CONDITIONS: Non Small Cell Lung Cancer; Small-cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — Fingolimod Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Efficacy in NSCLC (Experimental): n=22 NSCLC Any adult patients with lung cancer progressed on 2L+ systemic therapy n=any eligible patients from safety lead-in
  Interventions: Drug: Fingolimod 0.5 milligram (mg) [Gilenya]
- Efficacy in SCLC (Experimental): n=16 SCLC Any adult patients with lung cancer progressed on 2L+ systemic therapy n=any eligible patients from safety lead-in
  Interventions: Drug: Fingolimod 0.5 milligram (mg) [Gilenya]

INTERVENTIONS:
Drug: Fingolimod 0.5 milligram (mg) [Gilenya] — Oral fingolimod will be administered at a dose of 0.5 mg once a day.

SUMMARY:
This is a single-institution, open-labeled study using fingolimod (FTY720/Gilenya) in patients with non-small cell lung cancer (NSCLC) and small cell lung cancer (SCLC) who have progressed on chemo-immunotherapy. The study design will be a 6 patient safety lead-in with 2 cohorts of patients for efficacy analysis where fingolimod 0.5 mg will be taken orally once daily.

DETAILED DESCRIPTION:
Lung cancer is the second most common cancer and the leading cause of cancer death in the United States. There were approximately 237,000 new cases of lung cancer that were diagnosed in 2022 . The past decade has seen a revolution of new advances in the management of both non-small cell lung cancer (NSCLC) and small cell lung cancer (SCLC) with remarkable progress in screening, diagnosis, and treatment. The advances in systemic treatment have been driven primarily by the development of molecularly targeted therapeutics, immune-checkpoint inhibitors, and anti-angiogenic agents, all of which have transformed this field with significantly improved patient outcomes. Despite these advances, the prognosis for patients with advanced NSCLC and SCLC is poor, particularly after the failure of a platinum-based chemotherapy regimen and check point inhibitors with limited options available for patients. Therefore, new methods of targeting these malignancies are crucial. Fingolimod is a sphingosine analog that has demonstrated strong tumor suppressive activity in preclinical models of lung cancers and warrants further study.

This proposed study is a single institution Phase II clinical trial to investigate the safety and efficacy of fingolimod in patients with NSCLC and SCLC. Fingolimod is a small molecule derived from myriocin that acts as a sphingosine analog. It is currently FDA-approved to treat patients with relapsing forms of multiple sclerosis (MS), including clinically isolated syndrome, relapsing-remitting disease, and active secondary progressive disease by binding to sphingosine-1-phosphate (S1P) receptors 1, 3, 4, and 5 causing T lymphocyte egression and retention in peripheral lymphoid organs leading to immunosuppression. However, it can act as an antagonist for the S1P receptor promoting tumor suppression in multiple cancer cell lines and mouse models inhibiting cell proliferation, and inducing cancer cell death. There are multiple studies demonstrating its activity in preclinical models of lung cancer. Fingolimod induces a type of programmed cell death called necroptosis in lung cancer cells. This is mediated by activation of the tumor suppressor protein phosphatase 2A (PP2A) through interaction with the PP2A inhibitor (I2PP2A). Specifically, work done using the adenocarcinoma cell line A549 and small cell carcinoma cell line H1341 showed that fingolimod-mediated stress induced the formation of ceramidosomes leading to plasma membrane blebbing, compromised membrane integrity, and necroptosis.

This study will evaluate the safety, tolerability, and response rate in patients with NCSLC and SCLC who have progressed on front-line therapy including chemotherapy, immune checkpoint inhibitors, and targeted agents. It will contribute to the development of new methods for targeting these malignancies and provide insights into the potential use of fingolimod as a treatment option for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary, signed, and dated, Institutional Review Board (IRB) approved consent form in accordance with regulatory and institutional guidelines.
* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Male or female
* 18 years of age or older
* Measurable/evaluable as defined by RECIST 1.1 at baseline of advanced/metastatic non-small cell lung cancer progressed on 2L+ systemic therapy with any molecular subtype and PD-L1 Tumor Proportion Score (TPS).
* Measurable/evaluable as defined by RECIST 1.1 at baseline of extensive stage small cell lung cancer progressed on 2L+ systemic therapy.
* Ability to take oral medication and be willing to adhere to the fingolimod regimen.
* ECOG performance status 0-2
* Baseline lymphocyte count >1000 cells/mL
* For females of reproductive potential: use of highly effective contraception for at least 1 month before screening and agreement to use such a method during study participation and for an additional 2 months after the end of fingolimod administration.
* For males of reproductive potential: use of condoms or other methods during and for an additional 2 months after the end of fingolimod treatment to ensure effective contraception with a partner.

Exclusion Criteria:

* Patients who have had a recent (within the last 6 months) occurrence of cardiac event including myocardial infarction, unstable angina, stroke, transient ischemic attack, decompensated heart failure requiring hospitalization, or New York Heart Association Class III or IV heart failure, and congenital long QT-syndrome
* Patients who are receiving any medication(s) identified as having a Category D or higher interaction with the identified study agent who cannot be switched to another agent or discontinued before treatment if clinically appropriate. This medication review will be conducted by an oncology-trained Doctor of Pharmacy and discussed with the investigators before starting the treatment phase of this study. Careful evaluation for the following class of medications should be warranted due to their potential for severe side effects:
* Concurrent therapy with QT-prolonging medications with a known risk of torsade de pointes
* Concurrent therapy with drugs that slow heart rate or atrioventricular conduction
* Concurrent therapy with antineoplastic, immunosuppressive, or immune-modulating therapies
* Patients taking ketoconazole who have not completed their last dose at least 2 weeks before starting fingolimod.
* Active untreated brain metastases. Patients are eligible if brain metastases are previously treated and are asymptomatic. Patients must be neurologically stable and must be on stable or tapering corticosteroids 2 weeks before Cycle 1 Day 1
* Patients who have a history or presence of Mobitz Type II 2nd-degree or 3rd-degree atrioventricular block or sick sinus syndrome, unless patients have a functioning pacemaker.
* Patients who have a baseline QTc interval ≥ 500 msec
* Patients who have cardiac arrhythmias requiring Class IA or Class III anti-arrhythmic drugs.
* Class IA: disopyramide (Norpace), quinidine (Quinidex), procainamide (Procanbid)
* Class III: dronedarone (Multaq), dofetilide (Tikosyn), sotalol (Betapace), ibutilide (Corvert), amiodarone (Nexterone)
* Patients who have a hypersensitivity or allergic reaction (including rash, urticaria, and angioedema) to fingolimod or any of the excipients.
* Patients who have an active, uncontrolled acute or chronic bacterial, viral, or fungal infection
* Patients who have not completed all immunizations in accordance with current immunization guidelines before initiating fingolimod therapy
* Unwillingness or inability to comply with procedures required in this protocol.
* Patients who are currently participating in any other clinical trial of an investigational product
* Female patients who are of child-bearing potential (WOCBP) who are pregnant, planning to become pregnant during the study, or lactating. A urine pregnancy test for WOCBP will be collected during the screening period. Females will be determined to be not of child-bearing potential with a history of hysterectomy, tubal ligation, or age 45 or older with postmenopausal status > 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Safety of Fingolimod | 6 months
  Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0.
Response Rate | 6 months
  To evaluate the objective response rate (ORR) (when measurable) according to RECIST 1.1 criteria

SECONDARY OUTCOMES:
Progression-free Survival | 6 months
  Progression-free survival (PFS) as measured from the date of the first study treatment to the date of the first objective documentation of radiographic disease progression or death due to any cause
Overall Survival | 6 months
  Overall survival (OS) as measured from the date of first study treatment to the date of death due to any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No